CLINICAL TRIAL: NCT06419543
Title: Paradoxical Reactions of Remimazolam in Pediatric Painless Gastrointestinal Endoscopy: Incidence, Characters and Its Impact on Prognostic Outcomes-- a Randomized, Controlled Clinical Trial
Brief Title: Paradoxical Reactions of Remimazolam in Pediatric Painless Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRPG
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Endoscopy, Gastrointestinal
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group R1 (Experimental): The first induction dose of remimazolam is 0.1mg/kg.
  Interventions: Drug: Remimazolam
- Group R2 (Experimental): The first induction dose of remimazolam is 0.2mg/kg.
  Interventions: Drug: Remimazolam
- Group R3 (Experimental): The first induction dose of remimazolam is 0.3mg/kg.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Observe the incidence of paradoxical reactions after the first induction.
  Other Names: remimazolam besylate

SUMMARY:
Exploring the effect of remimazolam dose on paradoxical reactions in pediatric painless gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Exploring the effect of remimazolam dose on paradoxical reactions and sedation in pediatric painless gastrointestinal endoscopy, observing the performance and duration of paradoxical reactions, and analyze the factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-12 years old
* ASA I-II level
* Sign an informed consent form

Exclusion Criteria:

* Developmental delay or neurological and psychiatric disorders
* Severe malnutrition or severe obesity
* High risk of stomach fullness and reflux aspiration
* Allergic to benzodiazepines and opioids
* Those who have taken sedative, analgesic, or antidepressant drugs within 24hours
* Severe sleep apnea
* Abnormal liver and kidney function
* Recently participated in other clinical studies

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
incidence of paradoxical reaction | 2 minutes after first infusion of remimazolam
  observe the incidence of paradoxical reaction within 2 minutes

SECONDARY OUTCOMES:
performance and duration of paradoxical reaction | 2 minutes after first infusion of remimazolam
  observe the performance and duration of paradoxical reaction within 2 minutes
dosage of sedative drugs | First infusion until end of remimazolam administration
  Total dose of the first administered plus supplemental doses of sedative drugs.
time records | 1 day
  anesthesia time, induction time, surgical time, awakening time, and recovery time
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 day
  respiratory suppression incidence;intraoperative blood pressure and heart rate changes: record the patient's intraoperative blood pressure, heart rate, and the use of related vasoactive drugs; postoperative adverse reactions: such as hypertension, hypotension, tachycardia, gastrointestinal symptoms, postoperative restlessness, etc.

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospita
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No